CLINICAL TRIAL: NCT07000422
Title: Effect of Eye Movement Exercise on Gait Spatial and Temporal Parameters in Cerebral Palsy Spastic Diplegic Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salma Mohammed Hamza Rizq, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004463
Record Dates: First submitted 2025-05-24; First posted 2025-06-02 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Palsy Spastic Diplegia
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selected gait training program (Active Comparator): They will receive selected gait training (treadmill) sessions for five times per week over 6 successive months.
  Interventions: Other: Selected gait training program
- Selected gait training program + Eye movement exercise (Experimental): They will receive selected gait training (treadmill) sessions plus eye movement exercise for five times per week over 6 successive months.
  Interventions: Other: Selected gait training program; Other: Eye movement exercise

INTERVENTIONS:
Other: Selected gait training program — All children in both groups will receive selected gait training (treadmill) sessions for five times per week over 6 successive months.
Other: Eye movement exercise — All children in the experimental group will receive eye training exercises for five times per week over 6 successive months. The exercises include tasks to improve visual focus and tracking. Children search for a specific card among 20 while covering one eye, repeated 10 times. They follow a pencil moving vertically, horizontally, in circles, and in a figure 8, maintaining a 1m distance. Exercises include shifting gaze between two pencils, recognizing letters on a shaking card, and tracking a pencil from 5cm to 50cm. Tasks are done with each eye covered separately. Another task involves walking while focusing on a fixed target 1m away at eye level for 5 minutes.
  Arms: Selected gait training program + Eye movement exercise

SUMMARY:
The purpose of this study is to determine if there is an effect of eye movement training exercises on gait kinetic variables in cerebral palsy spastic diplegic children.

DETAILED DESCRIPTION:
Cerebral palsy is often accompanied by a dysfunction of the visual system consisting of an anterior part both eyes and the optic nerves up to the optic chiasm and a posterior part--the optic tracts, the lateral geniculate nuclei, the optic radiations and the occipital cortex. among children with cerebral palsy, 49.6% had ophthalmological disorders. The eye movement disorders are most common showing functional abnormalities such as gaze, saccade, and smooth pursuit in addition to strabismus and abnormal eye movements. In other words, the aspects of cerebral palsy are based not only on motor dysfunction characteristics and local anatomy but also on neuro-ophthalmology.

The visual perception system has a great influence on postural control and motor development by engaging in spatial association, identifying object characteristics, and distinguishing objects and their backgrounds, and eye movement function to place the image of nearby objects in the center also acts as an important factor in postural control and motor development. Eye movement control is the most basic type of visual perception, and lack of eye movement control often occurs in patients suffering from central nervous system diseases.

In order to achieve balance during normal gait, diverse brain regions, such as the cerebral cortex, cerebellum, and brain stem are involved. There are three crucial functional factors: the supporting action of the musculoskeletal system, the coordination of functional eye movement, and the integration of sensory function with action.

Eye movement training, in which movement patterns are adjusted through visual feedback, has been studied recently. Visual field and visual accuracy affect balance and movement ability, and in particular, patients with problems in the visual system often develop problems with balance ability.

The vestibular system contributes to postural stability and visual stabilization through the vestibulo-spinal reflex (VSR) and the vestibulo-ocular reflex (VOR). The vestibulo-ocular reflex is a reflex eye movement that stabilizes images on the retina during head movement. A rotation of the head is detected, which triggers an inhibitory signal to the extraocular muscles on one side and an excitatory signal to the muscles on the other side. The result is a compensatory movement of the eyes. the vestibulo-ocular reflex does not depend on visual input and works even in total darkness or when the eyes are closed.

There is lack in research regarding the area improve eye ex. Its effect on motor ability as in gait, most eye movement studies have been focused on balance, and studies relating eye movement training to gait have been insufficient, so this study will be conducted in hope evidence this area.

ELIGIBILITY:
Inclusion Criteria:

* Their age range 4-6 years old.
* They are Classified on levels I and II of the Gross Motor Function Classification System (GMFCS).
* The degree of spasticity will range from grade 1 or 1+ according to Modified Ashworth Scale.
* They able to walk without the assistance of another individual.
* Children with spastic diplegia gait pattern of Crouch gait.
* Intact vision and clear eye investigations.
* They Able to follow the verbal command.

Exclusion Criteria:

* Orthopedic deformities, a history of surgery.
* A history of eye surgery, squint or optic neuropathy.
* Diagnosis of epilepsy or having experienced convulsive crises (whether treated with medication or not).

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-07 (Estimated)

PRIMARY OUTCOMES:
Step Length | 6 months
  Using the foot print, the distance from the heel of one foot-strike to the heel of the opposite foot-strike will be measured in centimeters before and after treatment for all participants in both groups.
Step Width | 6 months
  Using the foot print, the distance between the centers of the feet during the double limb support portion of the gait cycle will be measured in centimeters before and after treatment for all participants in both groups.
Stride Length | 6 months
  Using the foot print, the distance between heels of two consecutive foot-strikes of the same foot (distance of a whole gait cycle) will be measured in centimeters before and after treatment for all participants in both groups.
Cadence | 6 months
  Using the foot print, the number of steps per minute will be measured before and after treatment for all participants in both groups.
Step Time (s) | 6 months
  Using the foot print, the time elapsed from initial contact of one foot to initial contact of the opposite foot will be calculated in seconds before and after treatment for all participants in both groups.
Stride Time | 6 months
  Using the foot print, the time of one whole gait cycle (right foot hitting the ground, left foot hitting the ground, then right foot hitting the ground again) will be calculated in seconds before and after treatment for all participants in both groups.
Stance Time Stance Time | 6 months
  Using the foot print, the time from heel strike to toe off on the same foot will be calculated in seconds before and after treatment for all participants in both groups.
Swing Time | 6 months
  Using the foot print, the time from toe off to heel strike on the same foot will be calculated in seconds before and after treatment for all participants in both groups.
Single Support Time | 6 months
  Using the foot print, the time in one gait cycle in which only one foot is on the ground will be calculated in seconds before and after treatment for all participants in both groups.
Double Support Time | 6 months
  Using the foot print, the time in one gait cycle in which both feet are on the ground will be calculated in seconds before and after treatment for all participants in both groups.

SECONDARY OUTCOMES:
Ocular motor score (OMS) | 6 months
  It will be assessed for all participants in both group before and after treatment. It is a new clinical test protocol for evaluating ocular motor functions in children and young adults. OMS is a set of 15 important and relevant non-invasive ocular motor function parameters derived from clinical practice. The subtests are scored as 0 (normal) 0.3 or 0.5 (subnormal) and 1 (pathological).

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Elsayed mohamed Shoukry, PhD, Study Chair — Professor, Cairo university; Asmaa Osama Sayed, PhD, Study Director — Assistant Professor, Cairo university
Locations (1):
- Cairo University, Giza, Egypt